CLINICAL TRIAL: NCT01929538
Title: Covered Self-expandable Metal Stent, 6 Versus 12 Months, for Benign Biliary Stricture Caused by Chronic Pancreatitis: a Prospective Randomized Study
Brief Title: Covered Metal Stent for Benign Biliary Stricture Caused by Chronic Pancreatitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Leena Kylanpaa, MD, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 175/13/03/02/2013
Record Dates: First submitted 2013-08-14; First posted 2013-08-28 (Estimated); Last update posted 2022-08-17 (Actual); Status verified 2022-08

CONDITIONS: Biliary Stricture; Chronic Pancreatitis
Keywords: Chronic pancreatitis; Biliary stricture; Endoscopic treatment; cSEMS
MeSH Terms: conditions — Pancreatitis, Chronic | interventions — Cholangiopancreatography, Endoscopic Retrograde

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Covered biliary metal stent, 12 mm (Active Comparator): ERCP and placement of a covered self-expanding biliary metal stent, 12mm in diameter
  Interventions: Procedure: ERCP; Device: covered self-expanding biliary metal stent, 12mm in diameter
- covered Biliary metal stent, 10 mm (Active Comparator): ERCP and placement of a covered self-expanding biliary metal stent, 10 mm in diameter
  Interventions: Procedure: ERCP; Device: covered self-expanding biliary metal stent, 10mm in diameter

INTERVENTIONS:
Procedure: ERCP — endoscopic retrograde cholangiopancreatography
Device: covered self-expanding biliary metal stent, 12mm in diameter
  Arms: Covered biliary metal stent, 12 mm
Device: covered self-expanding biliary metal stent, 10mm in diameter
  Arms: covered Biliary metal stent, 10 mm

SUMMARY:
Benign biliary strictures caused by chronic pancreatitis can be endoscopically treated with covered self-expandable metal stents (cSEMS).The purpose of the prospective randomized study is to define the optimal duration of stenting and the diameter of the cSEMS.

DETAILED DESCRIPTION:
All consecutive patients admitted for ERCP and treated for benign biliary stricture caused by chronic pancreatitis with or without acute pancreatitis are prospectively enrolled in the study. The age and gender of the patients and the aetiology of the pancreatitis will be recorded.

At initial presentation, clinical and laboratory findings recorded include liver function tests, abdominal pain, jaundice and cholangitis. Pancreatic calcifications are documented in abdominal computed tomography. Patients with malignancies, cirrhosis, acute/chronic hepatitis or abnormal hepatic imaging studies are excluded. Patients with first attack of acute pancreatitis will be excluded.

The approval of the ethics committee of the hospital has been obtained. An informed consent will be obtained from all patients.

All patients are prepared and sedated for ERCP as per standard medical practice of the hospital. At the initial ERCP, an endoscopic sphincterotomy will be performed and the presence/absence of bile duct stones above the stricture and the treatment of stones are recorded. A pancreatic stent will be inserted if indicated. For the initial ERCP the patients will be randomized into two groups: those who receive 10 mm diameter cSEMS and those who receive 12 mm diameter cSEMS into the bile duct. For the randomization, sealed envelopes will be used. The length of the cSEMS is recorded.

Further ERCP for stent removal will be performed after six months for the patients with 12 mm diameter cSEMS and after twelve months for the patients with 10 mm diameter cSEMS. In case of stent migration during the follow-up, the stent will be replaced by a similar new cSEMS. If a pancreatic stent will be placed, the removal or replacement will be handled according to the hospital practice.

After each ERCP procedure, all patients will stay in hospital for monitoring the occurrence of primary complications such as acute pancreatitis and cholangitis, bile leak, bleeding or perforation. Plasma amylase activity is measured same day > 4h after ERCP. Post-ERCP pancreatitis is defined as the presence of abdominal pain attributable to acute pancreatitis and plasma amylase level at least three times above the upper limit of the reference interval. The treatment of primary complications is recorded.

Follow-up

Clinical response (adequate biliary drainage) and recurrent stricture formation are the primary endpoints of the study. Therefore, blood liver function tests (bilirubin, alkaline phosphatase) as well as the minimum diameter of the common bile duct in the area of the stricture, the maximum diameter of the common bile duct above the stricture and the length of the stricture are measured at ERCPs at the time of the initial ERCP and at removal of cSEMS. Blood liver function tests are measured in the morning before ERCPs; the exact widths and lengths in mm:s are obtained by comparison the widths and lengths with the diameter of the scope. In addition, blood liver function tests are measured and abdominal ultrasonography performed in the follow-up six months and two years after the stent removal.

Morbidity and mortality are additional endpoints of the study. Therefore, complications (deaths, stent occlusions, dislodgements or migrations, cholangitis, hemobilia, stone formation above the stent), management of complications, admission times, surgical interventions and any additional care needed are monitored and recorded during the follow-up time. Patients are asked to contact the physician at any time if symptoms such as fever, abdominal pain or jaundice occur.

ELIGIBILITY:
Inclusion Criteria:

* Benign biliary stricture caused by chronic pancreatitis

Exclusion Criteria:

* Malignancy, cirrhosis, acute/chronic hepatitis or abnormal hepatic imaging. First attack of acute pancreatitis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2013-08; Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Stricture resolution of the common bile duct in the two study groups | 2,5 years
  Stricture resolution during stenting and follow-up period, defined by normal liver function tests and abdominal ultrasonography

SECONDARY OUTCOMES:
Stent removability | 1 year
  Ability to remove stents endoscopically after six months and one year without stent-removal related complications
Occurrence of complications related to stents and procedure | 2,5 years

OTHER OUTCOMES:
Biliary stricture Chronic pancreatitis | 2,5 years

CONTACTS AND LOCATIONS:
Overall Officials: Leena Kylänpää, MD, PhD, Principal Investigator — Helsinki University Central Hospital
Locations (1):
- Helsinki University Central Hospital, Helsinki, Finland